CLINICAL TRIAL: NCT00003637
Title: Standard Radiotherapy Versus Concurrent Chemo-Radiotherapy Followed by Adjuvant Chemotherapy for Locally Advanced (Non-Metastatic) Nasopharyngeal Cancer
Brief Title: Radiation Therapy Alone Compared to Radiation Therapy Plus Chemotherapy in Treating Patients With Previously Untreated Cancer of the Nasopharynx
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066722; NMRC-SQNP01; EU-98047
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-01

CONDITIONS: Head and Neck Cancer
Keywords: stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Fluorouracil; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether radiation therapy alone is more effective than radiation therapy plus chemotherapy in treating cancer of the nasopharynx.

PURPOSE: This randomized phase III trial is studying how well radiation therapy and chemotherapy works compared to radiation therapy alone in treating patients with previously untreated cancer of the nasopharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the clinical response, distant metastases, disease-free survival, and overall survival in patients with previously untreated, locally advanced, nonmetastatic nasopharyngeal cancer treated with radiotherapy alone vs concurrent chemoradiotherapy followed by adjuvant chemotherapy.

OUTLINE: This is a randomized study.

Patients are randomized to receive radiotherapy alone (arm I) or concurrent chemoradiotherapy followed by adjuvant chemotherapy (arm II).

* Arm I: Patients receive radiotherapy once daily 5 times a week for 7 weeks.
* Arm II: Patients receive cisplatin IV over 6-8 hours for 4 consecutive days every 3 weeks for 3 courses. Concurrent radiotherapy is given once daily 5 times a week over the 7 week treatment period. This chemoradiotherapy is followed 3 weeks later by adjuvant chemotherapy. Patients receive cisplatin IV and fluorouracil IV over 6-8 hours for 4 consecutive days every 4 weeks for 3 courses.

Patients are followed every 4 months for the first year, every 6 months for the next 2 years, and then annually thereafter until death.

PROJECTED ACCRUAL: A minimum of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nasopharyngeal cancer that is previously untreated WHO Type III
* Stage III/IV (T3-4 Nx M0 or Tx N2-3 M0) confirmed by CT PNS
* No evidence of distant metastases detected on chest x-ray, bone scan, and liver ultrasound

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* SAP and SGOT less than 2 times upper limit of normal
* Bilirubin less than 1.4 mg/dL

Renal:

* Creatinine less than 1.6 mg/dL
* Creatinine clearance greater than 50 mL/min

Other:

* No other malignant disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* See Disease Characteristics
* No concurrent aminoglycoside antibiotics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1998-09

PRIMARY OUTCOMES:
Clinical response
Distant metastases
Disease-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Eu J. Chua, MD, Study Chair — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore